CLINICAL TRIAL: NCT05316571
Title: Sitting Interruption and Whole-body Cardiovascular Health: Linking Physiological Responses to Risk Behaviors
Brief Title: Sitting Interruption and Whole-body Cardiovascular Health
Acronym: SWITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-3195; 1R01HL157187-01A1 (NIH)
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sedentary Behavior; Sedentary Time
Keywords: Sedentary Behavior; Interruption; Sitting; Cardiovascular; Arterial Stiffness; Pulse Wave Velocity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Each participant will complete four, 4-hour SB bouts with the following conditions: (i) one 5-minute walk break per hour; (ii) one 15-minute standing break per hour; (iii) two breaks per hour, alternating between 5 minutes of walking and 15 minutes of standing; and (iv) SB with no breaks (control). The order of intervention will be assigned in a randomized, crossover manner with 24 potential unique sequences of intervention assignment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers and participants will be blinded to the condition until each day of testing, and the statistician and any technicians processing outcome data will be blinded to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One 5-Minute Walking Bout Each Hour (Active Comparator): A 4-hour sedentary behavior bout, during which the participant remains seated while watching a non-stimulatory documentary.
  The interruption strategy includes breaking up the 4-hour sitting bout with one 5-minute light intensity walking bout each hour. Each participant will be re-randomized to any of the non-completed arms after completion of the initial 4-hour sitting bout and interruption strategy until all arms have been completed.
  Interventions: Behavioral: One 5-Minute Walking Bout Each Hour
- One 15-Minute Standing Bout Each Hour (Active Comparator): A 4-hour sedentary behavior bout, during which the participant remains seated while watching a non-stimulatory documentary.
  The interruption strategy includes breaking up the 4-hour sitting bout with one 15-minute standing bout each hour. Each participant will be re-randomized to any of the non-completed arms after completion of the initial 4-hour sitting bout and interruption strategy until all arms have been completed.
  Interventions: Behavioral: One 15-Minute Standing Bout Each Hour
- One 5-Minute Walking Bout and One 15-Minute Standing Bout Each Hour (Active Comparator): A 4-hour sedentary behavior bout, during which the participant remains seated while watching a non-stimulatory documentary.
  The interruption strategy includes breaking up the 4-hour sitting bout with one 5-minute light intensity walking bout and one 15-minute standing bout each hour. Each participant will be re-randomized to any of the non-completed arms after completion of the initial 4-hour sitting bout and interruption strategy until all arms have been completed.
  Interventions: Behavioral: One 5-Minute Walking Bout and One 15-Minute Standing Bout Each Hour
- Uninterrupted Sitting (Active Comparator): A 4-hour sedentary behavior bout, during which the participant remains seated while watching a non-stimulatory documentary.
  This uninterrupted sedentary bout will serve as a control. Each participant will be re-randomized to any of the non-completed arms after completion of the initial 4-hour sitting bout and interruption strategy until all arms have been completed.
  Interventions: Behavioral: Uninterrupted Sitting

INTERVENTIONS:
Behavioral: One 5-Minute Walking Bout Each Hour — One 5-minute light intensity walking break per hour throughout the 4-hour SB condition
  Arms: One 5-Minute Walking Bout Each Hour
Behavioral: One 15-Minute Standing Bout Each Hour — One 15-minute standing break per hour throughout the 4-hour SB condition
  Arms: One 15-Minute Standing Bout Each Hour
Behavioral: One 5-Minute Walking Bout and One 15-Minute Standing Bout Each Hour — Two breaks per hour throughout the 4-hour SB condition, alternating between a 5-minute light intensity walking break and a 15-minute standing break
  Arms: One 5-Minute Walking Bout and One 15-Minute Standing Bout Each Hour
Behavioral: Uninterrupted Sitting — No breaks will be provided throughout the 4-hour SB condition. This will be used as the control condition
  Arms: Uninterrupted Sitting

SUMMARY:
There is strong evidence for the association between sedentary behaviors and cardiovascular diseases such as coronary heart disease and stroke. However, the public currently has no clear guidance on how to limit or interrupt their sedentary behaviors. This study will identify and test the physiological effects of several sedentary behavior interruption strategies and explore the feasibility (i.e., likelihood of an individual performing the requested activities) of those strategies to inform the development of public policy surrounding sedentary behavior interruption. Long-term, the findings of this study will inform a large clinical trial that can test whether sedentary behavior reduction can decrease cardiovascular disease risk.

DETAILED DESCRIPTION:
Sedentary behaviors (SB) are biologically distinct but understudied heart disease risk factors. National and international agencies have concluded that the level of evidence for an overall and dose-response association between SB and heart disease mortality is moderate-strong. These agencies do not provide specific recommendations for breaking-up SB, though do call on the research community to facilitate policy development by establishing biological plausibility, identifying the optimal dose for SB substitution strategies, and conducting randomized clinical trials to test the efficacy of these strategies. Accordingly, the goal of this study is to identify mechanism-informed, socioecological-based SB substitution recommendations to reduce heart disease risk. To achieve this goal, two aims will be addressed. Aim 1 will identify a feasible SB substitution strategy to prevent the negative cardiovascular responses to prolonged SB (i.e., strategies that people will actually follow). Adverse cardiovascular responses to prolonged SB will be measured using aortic arterial stiffness (AS), a noninvasive test that predicts future heart disease. To accomplish this aim, 56 middle-aged (30-60 years) participants will provide written informed consent, prior to the measurement of aortic AS and associated mechanistic responses to the following over 4 hours, in a randomized crossover manner: (i) SB with a 5-minute walk break once per hour; (ii) SB with a 15-minute standing break once per hour; (iii) SB with two breaks per hour, alternating between a 5-minute walk and a 15-minute stand; and (iv) SB with no breaks (control). These strategies were selected based on extensive prior work by the investigators, and because they are feasible, which is a key component of this study. SB reduction strategies will only decrease heart disease risk if people are willing to adhere to future SB substitution recommendations. To increase the likelihood of feasibility and long-term adherence, Aim 2 will evaluate the determinants of SB using a socioecological model. This recognizes that behavior change is likely to be limited if the physical and sociocultural environments do not support the behavior change. To accomplish Aim 2, a combined inductive-deductive qualitative approach will be used. Participants who complete Aim 1 will participate in one of 6 focus groups (6-8 participants/group). Crucially, the outcomes from this proposal will be instrumental in helping to design a subsequent clinical trial to test a mechanism-informed yet feasible SB reduction intervention, and in doing so directly support the development of SB policy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30-60 years
* Insufficiently active: self-reported exercise <90 minutes per week for the past 3 months
* Sedentary: self-reported sitting >8 hours per day
* Self-reported ability to walk 4 blocks and climb 2 flights of stairs
* Possession of cellular phone able to receive text messages

Exclusion Criteria:

* Use of assisted-walking devices
* Comorbid condition that would limit the ability to reduce sedentary behavior (e.g., musculoskeletal condition, current chemotherapy)
* Plans for major surgery within next 3 months
* Recent history (<1 year) of ischemic heart disease, chronic heart failure, stroke, or chronic kidney disease
* Recent (< 1 year) or planned bariatric surgery
* Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg
* Current or recent (within last 6 months) pregnancy; current or recent (within last 3 months) breastfeeding
* Morbidly obesity (BMI >40 kg/m^2) or underweight (BMI <18.5 kg/m^2)
* Use of anti-hypertensive drugs
* Use of glucose-controlling medication
* Heavy alcohol consumption (>15 drinks per week)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Carotid-femoral Pulse Wave Velocity (cfPWV) | Measurements will be taken immediately before and after each 4-hour SB condition
  cfPWV (m/sec) will be measured between the carotid and femoral arteries, using a collar around the neck and a cuff around the thigh, with the participant in a supine position. cfPWV is calculated by dividing path length by pulse transit time and reported as the mean of three measurements

SECONDARY OUTCOMES:
Change in Heart-middle Cerebral Artery Pulse Wave Velocity (Brain PWV) | Measurements will occur continuously throughout each of the 4-hour SB conditions
  Brain PWV (cm/sec) is the velocity at which a pressure wave travels between the heart and cerebrovascular system. Brain PWV will be calculated from the ECG r-wave to the foot of the Cerebral Blood Flow Velocity (CBFV) waveform
Mean Change in Femoral-ankle PWV | Measurements will be taken immediately before and after each 4-hour SB condition
  Femoral-ankle PWV (m/sec) is the velocity at which a pressure wave travels between the femoral-ankle arterial segments. Femoral-ankle PWV is calculated by dividing path length by pulse transit time and reported as the mean of three measurements

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hanson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months following publication and continuing for 36 months
Access Criteria: Investigator has IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Higgins S, Cowley ES, Paterson C, Hanson ED, Dave GJ, Meyer ML, Lin FC, Gibbs BB, Vu M, Stoner L. Protocol for a study on Sitting with Interruption and Whole-Body Cardiovascular Health (SWITCH) in middle-aged adults. Contemp Clin Trials. 2023 Feb;125:107048. doi: 10.1016/j.cct.2022.107048. Epub 2022 Dec 9. PMID 36509249